CLINICAL TRIAL: NCT05025930
Title: Evaluate the Safety and Effectiveness of the Endoscopic Surgical Instrument Control System (SP1000): a Multi-center, Randomized, Single-blind, Parallel Controlled Clinical Tria
Brief Title: Evaluate the Safety and Effectiveness of the Endoscopic Surgical Instrument Control System (SP1000).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Chinese PLA General Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Edge Medical Robotics CO.,LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SysMU-Robot
Record Dates: First submitted 2021-07-09; First posted 2021-08-30 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Urologic Neoplasms
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic surgical instrument control system (SP1000: single- port laparoscopy) (Experimental): Urological surgery procedures such as prostatectomy, and partial or radical nephrectomy will be performed using endoscopic surgical instrument control system (SP1000)
  Interventions: Device: endoscopic surgical instrument control system (SP1000: single-port laparoscopy)
- Comparator: endoscopic surgical instrument control system (IS3000: multi-port laparoscopy) (Active Comparator): Urological surgery procedures such as prostatectomy, and partial or radical nephrectomy will be performed using endoscopic surgical instrument control system (IS3000)
  Interventions: Device: endoscopic surgical instrument control system (IS3000: multi-port laparoscopy)

INTERVENTIONS:
Device: endoscopic surgical instrument control system (SP1000: single-port laparoscopy) — The system will be used in conjunction with other equipment during endoscopic surgery to accurately control endoscopic surgical instruments and perform delicate surgical procedures such as grasping, cutting, blunt separation, hemostasis, ligation and suture.
  Arms: endoscopic surgical instrument control system (SP1000: single- port laparoscopy)
Device: endoscopic surgical instrument control system (IS3000: multi-port laparoscopy) — The system will be used in conjunction with other equipment during endoscopic surgery to accurately control endoscopic surgical instruments and perform delicate surgical procedures such as grasping, cutting, blunt separation, hemostasis, ligation and suture.
  Arms: Comparator: endoscopic surgical instrument control system (IS3000: multi-port laparoscopy)

SUMMARY:
Robot-assisted surgery has been successfully adopted rapidly over the last decade. Robotic technology with tridimensional imaging can improve operating dexterity, visualization of difficult anatomic locations. This is a prospective study aims to evaluate the safety and effectiveness of the domestic surgical robot.

DETAILED DESCRIPTION:
In this clinical trial, the subjects will be randomly divided into two groups, and the urological typical surgical procedures (prostatectomy, and partial or radical nephrectomy) will be performed with the endoscopic surgical instrument control system SP1000 and IS3000.And the non-inferiorly comparison will be made between the surgical results of two systems to verify the safety and effectiveness of the endoscopic surgical instrument control system (SP1000).

ELIGIBILITY:
Inclusion Criteria:

1. Any male or female age from 18 to 80
2. BMI 18-30kg/m2
3. Have urological surgery indications (cystectomy, prostatectomy, and nephrectomy)
4. Patients with physiologic conditions capable of receiving laparoscopic surgery
5. Be able to cooperate and complete the follow-up and related examinations
6. Volunteer to participate in this study and sign the informed consen

Exclusion Criteria:

1. The researchers assess patients with severe cardiovascular or circulatory disease and cannot tolerate the surgery
2. History of epilepsy or mental illness
3. Pregnant and lactation
4. Surgery history at the relevant surgical site, which is considered to influence surgical procedures
5. Severe allergic or addiction of drug and alcohol
6. Abdominal infection, peritonitis, diaphragmatic hernia, severe systemic infection or metastasis disease
7. Inability to understand the trial or complete the follow-up
8. Participated in other therapeutic clinical trials within 90 days
9. Patients who had undergone major operation and major trauma within 28 days prior to enrollment, which the researchers considered to have an impact on the outcome of surgery
10. Patients deemed unsuitable to participate in this trial by researchers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Surgical success rate | 24 hours
  The surgical success rate was defined as the percentage of patients in the experimental group and the control group who were successfully operated with the systems
Incidence of serious adverse events during clinical trial | 3 months

SECONDARY OUTCOMES:
Perioperative complication rate | 3 months
  Perioperative complication will be graded using the Clavien-Dindo Complication Classification. The proportion and severity of perioperative complications will be analyzed
Changes in serum creatinine | 3 months
  Evaluating renal function by changes in serum creatinine after surgery for partial or radical nephrectomy
Changes in prostate-specific antigen levels | 3 months
  Changes in prostate-specific antigen levels will be measured after surgery for patients who undergone radical prostatectomy
Tumor recurrence rate | 3 months
Machine installation time | preoperative
  Time from sheeting to complete the installation of surgical instruments
Operative time | 12 hours
Blood loss during the surgery | 12 hours
Margin positive rate | 1 month
Pain after surgery | 24 hours
  Visual analogue scale as a monitoring tool for postoperative pain
Surgeon Satisfaction | 12 hours
  NASA-TLX quantification table will be used to evaluate surgeon satisfaction after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tianxin Lin, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No